CLINICAL TRIAL: NCT05921292
Title: A Clinical Study to Evaluate the Omeza Combination Therapy for the Management and Treatment of Chronic Cutaneous Wounds/Ulcers of Multiple Etiologies
Brief Title: Omeza Combination Therapy for the Management and Treatment of Chronic Cutaneous Wounds/Ulcers of Multiple Etiologies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Omeza, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OM-CTP-002
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Non-healing Wound; Non-Healing Ulcer of Skin
MeSH Terms: interventions — oncomodulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Omeza® Products Used in Combination (Experimental): Subjects in this single-arm study will have the targeted wound/ulcer treated with a combination therapy which includes the use of a wound preparation (2mL vial), a skin protectant (2mL vial), and a wound matrix (1.6g vial). Patients will be treated weekly for four weeks. Treatment may be continued weekly for an additional 8 weeks with participant and investigator agreement.
  Interventions: Combination Product: Omeza Products Used in Combination

INTERVENTIONS:
Combination Product: Omeza Products Used in Combination — Subjects in this single-arm study will have the targeted wound/ulcer treated with Omeza® combination therapy which includes the use of the following products:
  * Omeza® Lidocaine Lavage
  * Omeza® Complete Matrix (OCM™)
  * Omeza® Skin Protectant At each treatment (on days 0, 7, 14, 21; +/- 3 days each), the patient's intact skin around the wound/ulcer will be prepped with Omeza® Lidocaine Lavage. OCM™ will be applied directly to the wound/ulcer and Omeza® Skin Protectant will be applied to the periwound and surrounding intact skin. Treatments may be repeated during an optional 7 additional weeks (on days 28, 35, 42, 49, 56, 63, and 70; +/- 3 days each). Final assessment will be made at week 12.
  Other Names: Omeza® Lidocaine Lavage, Omeza® Complete Matrix (OCM™), and Omeza® Skin Protectant

SUMMARY:
The goal of this clinical trial is to evaluate the use of Omeza combination therapy with Standard of Care. The main question it aims to answer is:

- Can Omeza combination therapy with Standard of Care enable chronic wounds to begin a healing trajectory in a 4-week period?

Patients will be treated with:

* OCM™ Wound Matrix
* Omeza combination therapy
* Standard of Care

DETAILED DESCRIPTION:
The goal of this clinical trial is to demonstrate that the Omeza combination therapy with Standard of Care supports chronic wounds to move from chronicity to a healing trajectory. The trial is targeting those wounds that have failed therapy prior to trial enrollment and are chronic by definition of no change in area size after 2 weeks of standard of care treatment. The inclusion and exclusion criteria applied to this chronic wound clinical trial is broadened with the intention to include all patients and outliers that would not qualify for controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old and female subjects are not pregnant
* Willing and able to comply with Trial procedures, including Trial visits and Trial dressing regimens
* Targeted chronic wound/ulcer has been chronically present for at least two (2) months (8 weeks) as of the date the subject signs consent for study
* Study target chronic wound/ulcer size is a minimum of 2.0 cm2 and a maximum of 100.0 cm2 without exposed tendon, muscle or bone
* Willing and able to comply with study procedures, including study visits and study dressing regimens including ability of the subject to tolerate limb compression bandage, when applicable
* Subject has read and signed the IRB-approved Informed Consent Form before screening procedures are undertaken.

Additional Inclusion Criteria (for Subjects with Wounds/Ulcers in Lower Extremities):

* The affected limb must have adequate perfusion confirmed by vascular assessment. Any one of the following methods performed within 1 or 2 months of the first screening visit are acceptable:

  1. Ankle Brachial Index (ABI) between 0.8 and 1.3
  2. Toe Brachial Index (TBI) > 0.6
  3. Transcutaneous oximetry (TCOM) >40mmHg
  4. Pulse volume recording (PVR): biphasic or triphasic waveforms
* Confirmation of venous disease by non-invasive venous studies with either Doppler confirmed venous reflux or having ≥ 2 clinical characteristics of venous insufficiency (varicose veins, lipodermatosclerosis, venous dermatitis, atrophie blanche, edema). Biopsy done to exclude other skin conditions e.g., cancer on ulcers ≥ 6 months
* Have a venous ulcer between the knee and ankle, at or above the malleolus
* Subject understands and is willing to participate in the clinical study visits including compression if needed for minimum 14 days (compression dressing changed once weekly) prior to study start, participate in the informed consent process, and can comply with weekly visits and the follow-up regimen
* If more than one chronic wound/ulcer is present on the same leg, they must be greater than 2 cm apart and only the larger chronic wound/ulcer will be included in the study (i.e., targeted lesion)

Additional Inclusion Criteria (for Subjects with Diabetic Foot Ulcer):

* Diagnosed as having Type 1 or Type 2 diabetes
* Any lower extremity wound should have at least one method of arterial testing (ABI, TBI, Arterial Doppler with Waveforms, Pulse Volume Recordings, Skin Perfusion Pressure, TcPO2) within 1 or 2 months of the first screening visit.
* Presence of a DFU, Wagner 1 or 2 (see Appendix D for definitions), extending at least through the dermis provided it is below the level of the medial or lateral malleolus.
* Known HbA1c of ≤12% within 6 months
* The target wound will be located on the foot or ankle and will be the largest ulcer if two or more DFUs are present with the same Wagner grade and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 1 cm distant from the target wound

Exclusion Criteria:

* Targeted chronic wounds/ulcers exhibit clinical signs and symptoms of infection, as evidenced by tissue necrosis, redness, pain, and/or purulent drainage and/or receiving systemic antibiotics for the treatment of such*
* Targeted chronic wound/ulcer treated with a topical antibiotic within the last 7 days prior to first treatment with Omeza products.

  a. NOTE: washout of topical antibiotics and antibacterial treatments (eg. Silver, manuka honey, iodine, etc) is at least 7 days before first treatment with Omeza products.
* Targeted chronic wound/ulcer has been treated with any placental derived products, engineered material (e.g., Apligraf® or Dermagraft®) or other scaffold materials (e.g., Oasis, PuraPly AM or Matristem) within the last 30 days.
* Targeted chronic wound/ulcer requires enzymatic debridement during the study
* Targeted chronic wound/ulcer decreases in area by 30% or more during the 14 days screening/run-in period.
* Subjects who are unable to understand the aims and objectives of the trial or have a known history of poor adherence with medical treatment.
* Subject is medically unable to consent (due to head trauma, coma, etc.) or cognitively impaired (due to being mentally challenged, having Alzheimer's, etc.)
* Presence of any condition(s) that seriously compromises the subject's ability to complete this study.
* Subjects with a BMI>65
* Subject has any history of fish allergy or a known sensitivity to any of the SoC materials which contact the skin
* Presence of any monophasic waveforms on segmental Arterial Doppler/Pulse Volume Recording
* Subject is on dialysis
* Any active cancer other than a nonmelanoma skin cancer; any previous cancer must be in remission for at least 1 year: bone cancer of metastatic disease of the affected limb, or has had chemotherapy within the last 12 months
* Suspicion of malignancy within chronic wounds/ulcers: A biopsy must be performed for any wound that has been present for > 6 months and has not previously been biopsied. A biopsy should be performed regardless of duration of wound If a clinical suspicion of malignancy exists in the opinion of the Investigator.
* Life expectancy < 6 months
* Subject has received within 28 days of screening a treatment which is known to interfere with or affect the rate and quality of wound healing (e.g., thrombolysis, systemic steroids, immunosuppressive therapy, autoimmune disease therapy, dialysis, radiation therapy at wound site, chemotherapy) or who may receive such medications during the screening period or who has anticipated to require such medications during the course of the study at the discretion of the treatment PI.
* Untreated osteomyelitis
* Acute deep venous thrombosis
* Allergy to lidocaine and/or epinephrine
* Subject's inability to successfully tolerate compression therapy that is changed weekly
* All females of childbearing potential who are not using a highly effective method of birth control (failure rate less than 1% per year), such as implants, injectables, combined oral contraceptives, some IUDs, practice sexual abstinence or have a vasectomized partner.
* The use of the following treatments are prohibited within 30 days prior to randomized treatment and throughout the study:

  1. Heat lamps
  2. UV lights
  3. Whirlpool baths
  4. Hyperbaric oxygen
  5. Topical or local insulin administration

Additional Exclusion Criteria (for Subjects with Wounds/Ulcers in Lower Extremities):

* The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 1 or 2 months of the first screening visit are exclusionary:

  1. Ankle Brachial Index (ABI) less than 0.7 or greater than 1.3
  2. Toe Brachial Index (TBI) < 0.6
  3. Transcutaneous oximetry (TCOM) <40mmHg
* Suspicion of malignancy within VLU
* Acute deep venous thrombosis
* Study target chronic wound/ulcer extends more than 50% below the malleolus.

Additional Exclusion Criteria (for Subjects with Diabetic Foot Ulcer):

* Target wound deemed by the investigator to be caused by a medical condition other than diabetes or subject has wounds secondary to a disease other than diabetes (e.g. vasculitis, neoplasms, or hematological disorders)
* The affected limb of the diabetic subject must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 1 or 2 months of the first screening visit are exclusionary:

  1. Ankle Brachial Index (ABI) between 0.8 and <1.3
  2. Toe Brachial Index (TBI > 0.6
* The subject is unable to safely ambulate with the use of a study required offloading method
* Subject has unstable Charcot foot or Charcot with bone exposed that could inhibit wound healing
* Osteomyelitis or bone infection of the affected foot as verified by x-ray within 30 days prior to randomization. (In the event of an ambiguous diagnosis, the subject will not be enrolled)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Chronicity of Wound Healing | 4 weeks
  The proportion of subjects with a clinically significant improvement in Study Ulcer Exudate Assessments at 4 weeks compared to baseline assessment.
Change in Wound Area | 4 weeks
  Percent change in wound area at 4 weeks as measured by wound imaging software. Sub-characterization will include wounds with baseline area of greater than or less than 100㎟.
Wound Healing | 4 weeks
  The objective response rate (ORR) will be used to define effectiveness at 4 weeks. The ORR is defined as the proportion of subjects at 4 weeks that have had at least a 40% reduction in the area of the wound volume from Day 0 measurements measured by wound imaging software.
Wound Closure | 12 weeks
  Proportion of subjects that have had complete closure at or prior to 12 weeks of treatment.

SECONDARY OUTCOMES:
Improvement in Quality of Life | 12 weeks
  Change in the subject's Quality of Life (QoL). A numerical validated QoL scale (wound QoL Appendix F) specific for wound healing will be provided for participants to complete on a scheduled visit basis up to 12 weeks from Day 0.
Reported Pain Perception | 12 weeks
  Reported changes in pain perception will use a 10 cm Visual Analogue Scale and subjects will mark on the line from no pain to worst pain possible each scheduled visit.
Drainage/Exudate and Infection | 12 weeks
  Change in drainage/exudate and infection assessments. Drainage/exudate and infection assessment will be provided by the investigator in assessment of wounds at each week when changing dressings at each visit.
Enhanced Activities in Daily Living | 12 weeks
  Changes in the enhanced activities in daily living. Enhanced activities in daily living will be measured in an instrumental ADL scale at scheduled visits: the Barthel Index that measures the following criteria: chair/bed transfers, ambulation, ambulation/wheelchair, stair climbing, toilet transfers, bowel control, bladder control, bathing, dressing, personal hygiene, and feeding.
Time to Closure | 12 weeks
  This will be the time from Day 0 to the day that 100% or reepithelization without drainage or exudate has occurred. In addition, any wounds/ulcers that have not had complete closure by week 12 the maximum reported closure will be reported, and the data censored at 12 weeks.
Incidence of Healing | 12 weeks
  The proportion of subjects in which complete closure has occurred by Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Bell, DPM, Study Director — Omeza Holdings, Inc
Locations (1):
- Christus St. Vincent, Santa Fe, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No